CLINICAL TRIAL: NCT01431989
Title: Evaluation of Pharmaceutical Bioequivalence of Amoxicillin Trihydrate - Clamoxyl 500mg/5mL (Glaxo Wellcome Production.) in the Form Powder for Oral Suspension Versus Amoxil ® 500mg/5mL (GlaxoSmithKline Mexico SA) in the Form of Powder for Oral Suspension in Healthy Volunteers and Fasting, Using Techniques of Liquid Chromatography
Brief Title: Amoxicillin Bioequivalence Study Brazil - Fast
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 115954
Record Dates: First submitted 2011-09-08; First posted 2011-09-12 (Estimated); Results first posted 2012-02-07 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Infections, Bacterial
MeSH Terms: conditions — Bacterial Infections | interventions — Suspensions; Amoxicillin; Powders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test formulation (Active Comparator): Test product: Amoxicillin powder for oral suspension (Clamoxyl®) 500mg/5mL in Period 1; followed by 14-days washout period during which no medication was administered; followed by reference product: Amoxil® 500mg/5mL in Period 2.
  Interventions: Drug: Amoxicillin powder for oral suspension (Clamoxyl®) 500mg/5mL
- Reference formulation (Active Comparator): Reference product: Amoxil® 500mg/5mL powder for oral suspension in Period 1; followed by 14-days washout period during which no medication was administered; followed by test product: Amoxicillin powder for oral suspension (Clamoxyl®) 500mg/5mL in Period 2
  Interventions: Drug: Amoxil® 500mg/5mL powder for oral suspension

INTERVENTIONS:
Drug: Amoxicillin powder for oral suspension (Clamoxyl®) 500mg/5mL — Test formulation
  Arms: Test formulation
Drug: Amoxil® 500mg/5mL powder for oral suspension — Reference formulation
  Arms: Reference formulation

SUMMARY:
This study is prospective, open-label, randomized, crossover, single dose, with 02 treatments, 02 sequences and 02 periods. The volunteers received, in each period, the reference or the test formulation, according to the randomization list, under fasting conditions, in order to evaluate if the reference and test formulations are bioequivalent.

DETAILED DESCRIPTION:
This study is prospective, open-label, randomized, crossover, single dose, with 02 treatments, 02 sequences and 02 periods. The objective is to confirm if two formulations of Amoxicillin trihydrate, in the form powder for oral suspension, are bioequivalent. The test product is Amoxicillin trihydrate - Clamoxyl 500mg/5mL (Glaxo Wellcome Production.) in the form powder for oral suspension and reference product is Amoxil ® 500mg/5mL (GlaxoSmithKline Mexico SA) in the form of powder for oral suspension. Twenty eight healthy volunteers, of both genders, were evaluated. The volunteers received, in each period, the reference or the test formulation, according to the randomization list, under fasting conditions. In each period blood samples are collected in the following times: 0.00 (prior to administration of medication); 0.25; 0.50; 0.75; 1.00; 1.25; 1.50; 1.75; 2.00; 2.50; 3.00; 4.00; 5.00; 6.00; 8.00 (after administration of medication). The comparative bioavailability of the two formulations was evaluated based in statistical comparisons of relevant pharmacokinetic parameters, obtained from data of drug concentrations in blood.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years
* Body mass index between 18,5 and 25,0, can vary up to 15% for the upper limit (18,5 and 28,75)
* Good health conditions
* Obtain signed informed consent

Exclusion Criteria:

* Results of laboratory tests outside the normal limits, unless they are considered clinically irrelevant
* The volunteers who underwent surgery or who were hospitalized for any reason before the start of the study will be reviewed by the physician on admission in the study, observing a period of exclusion of 4 to 8 weeks
* Positive test for hepatitis B, hepatitis C or HIV in pre study evaluation
* Known hypersensitivity to the study drug or to compounds chemically related
* Use of experimental drug or participation in any clinical study within 6 months prior to study initiation
* Use of regular medication within 2 weeks prior to study initiation
* History of alcohol or drugs abuse or intake of alcohol within 24 hours prior to the period of confinement
* Consume of inductive drugs and/or enzymatic inhibitors (CYP450 - hepatic), that are toxic for the organism or presenting long half-life's elimination within 30 days prior to study initiation
* Use of MAO and serotonin reuptake inhibitors within 2 weeks prior to study initiation
* Volunteers with psychiatric or psychological illness unless they are considered clinically irrelevant by the investigator
* History or presence of hepatic, renal or gastrointestinal illness or other condition that interferes on drug's absorption, distribution, excretion or metabolism
* History of neurological, endocrine, pulmonary, hematologic, immune, brain, metabolic or cardiovascular illness
* Hypo or hypertension of any etiologic that needs pharmacologic treatment
* History or clinical case of myocardial infarction, angina and/or heart failure
* The volunteer donated or lost 450 mL or more of blood within the 3 months prior to the study initiation
* The volunteer has any condition that obstructs his/her participation in the study according the investigator's judgement
* Smoking
* Positive beta HCG exam for women
* Breastfeeding women
* Women making use of contraceptive medication

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2011-05-27 (Actual); Primary Completion 2011-06-11 (Actual); Study Completion 2011-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Goiânia, Goiás, Brazil

REFERENCES:
- See also: Results for study 115954 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115954?search=study&study_ids=115954#rs

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a prospective, open-label, randomized, crossover, single-dose study in which two different treatments (Test Product versus Reference Product) were administered in two sequences in two study periods. The objective was to confirm if two formulations of Amoxicillin trihydrate, in the form of powder for oral suspension, are bioequivalent.
Groups:
- Test Product in Period 1: Reference Product in Period 2: Test product, Amoxicillin (Clamoxyl) 500 milligrams (mg)/5 milliliter (mL) powder for oral suspension, in Period 1; followed by a 14-day washout period during which no medication was administered; followed by reference product, Amoxil 500 mg/5 mL powder for oral suspension, in Period 2
- Reference Product in Period 1: Test Product in Period 2: Reference product, Amoxil 500 mg/5 mL powder for oral suspension, in Period 1; followed by a 14-day washout period during which no medication was administered; followed by test product, Amoxicillin (Clamoxyl) 500 mg/5 mL powder for oral suspension, in Period 2
Period: Period 1
Arm/Group | Test Product in Period 1: Reference Product in Period 2 | Reference Product in Period 1: Test Product in Period 2
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: 14-Day Washout Period
Arm/Group | Test Product in Period 1: Reference Product in Period 2 | Reference Product in Period 1: Test Product in Period 2
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Test Product in Period 1: Reference Product in Period 2 | Reference Product in Period 1: Test Product in Period 2
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Participants Receiving Both Test and Reference Products: Participants receiving either test product, Amoxicillin (Clamoxyl) 500 mg/5 mL powder for oral suspension, in Period 1; followed by a 14-day washout period during which no medication was administered; followed by reference product, Amoxil 500 mg/5 mL powder for oral suspension, in Period 2 or reference product in Period 1 and test product inPeriod 2
Arm/Group | Participants Receiving Both Test and Reference Products
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.54 (7.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 14
Race/Ethnicity, Customized [Number; unit: participants]
  White | 10
  Black | 4
  Mulatto | 14

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve of Plasma Concentration of Drug From Time 0 (Zero) to t (Last Measurable Concentration) (AUC0-t)
Description: The area under the plot of plasma concentration of drug against time (non-compartmental method), after drug administration, is defined as the area under the curve (AUC). AUC0-t is calculated from time 0 (prior to administration of medication) to time t (the time of the last quantifiable concentration). AUC is of particular use in estimating the bioavailability of drugs, by measuring the extent of absorption. ng, nanograms; mL, milliliter.
Time Frame: Collection points (hours [hrs]): 0.00; 0.25; 0.50; 0.75; 1.00; 1.25; 1.50; 1.75; 2.00; 2.50; 3.00; 4.00; 5.00; 6.00; 8.00 evaluated in both periods (Day 1 of Period 1 [Day 1 of study]; Day 1 of Period 2 [Day 15 of study])
Population: Entire Study Population
Measure: Mean (Standard Deviation); unit: ng per hour per ml (ng*hr/mL)
Groups:
- Test Product: Test product, Amoxicillin (Clamoxyl) 500 mg/5 mL powder for oral suspension, received in either Period 1 or Period 2
- Reference Product: Reference product, Amoxil 500 mg/5 mL powder for oral suspension, received in either Period 1 or Period 2
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 28 | 28
ng per hour per ml (ng*hr/mL) | 36431.460 (6806.797) | 40426.451 (7279.259)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — Equivalence analysis. This is a bioequivalence study performed to support the register of Clamoxyl 500 mg/5 mL, according to the requirements of Brazilian Regulatory Agency - National Agency of Sanitary Surveillance (ANVISA); p = 0.0000, ANOVA; ANOVA model: 1) Fixed effects: Sequence, Period, and Formulation; 2) Random effects: Volunteer (Sequence) and Residual; Ratio Geometric mean T/R formulation = 90.03, 90% CI 2-sided [86.99 to 93.17], Standard Deviation 7.53 — The ratio between the geometric means of the test (T) and reference (R) formulations was calculated. Standard deviation intra subject was obtained

2. Primary Outcome: Maximum Observed Concentration of Drug Through Time (Cmax)
Description: Cmax is defined as the maximum or "peak" concentration of a drug observed after its administration. Cmax is one of the parameters of particular use in estimating the bioavailability of drugs, by measuring the total amount of drug absorbed. Measurement is obtained directly from the plasma concentration curve of the drug (non-compartmental method).
Time Frame: Collection points (hrs): 0.00; 0.25; 0.50; 0.75; 1.00; 1.25; 1.50; 1.75; 2.00; 2.50; 3.00; 4.00; 5.00; 6.00; 8.00 evaluated in both periods (Day 1 of Period 1 [Day 1 of study]; Day 1 of Period 2 [Day 15 of study])
Population: Entire Study Population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 28 | 28
ng/mL | 13615.929 (3886.864) | 15176.107 (3144.162)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0018, ANOVA; ANOVA model: 1) Fixed effects: Sequence, Period, and Formulation; 2) Random effects: Volunteer (Sequence) and Residual; Ratio Geometric mean T/R formulation = 87.93, 90% CI 2-sided [82.55 to 93.65], Standard Deviation 13.83 — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Area Under the Curve of Plasma Concentration of Drug From Time 0 (Zero) Extrapolated to Infinity (AUC0-inf)
Description: Measurement of AUC0-inf is obtained directly from the plasma concentration curve of drug against time (non-compartmental method). AUC0-inf is calculated from time 0 (prior to administration of medication) extrapolated to infinity, by using the formula AUC0-inf = AUC0-t + Clast/Kel, where Clast is the last measurable concentration, and Kel is the first-order rate constant associated with the terminal portion of the curve. AUC is of particular use in estimating the bioavailability of drugs, by measuring the extent of absorption.
Time Frame: Collection points (hrs):0.00; 0.25; 0.50; 0.75; 1.00; 1.25; 1.50; 1.75; 2.00; 2.50; 3.00; 4.00; 5.00; 6.00; 8.00 evaluated in both periods (Day 1 of Period 1[Day 1 of study]; Day 1 of Period 2 [Day 15 of study])
Population: Entire Study Population
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 28 | 28
ng*hr/mL | 36908.392 (6875.785) | 40977.755 (7372.809)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0000, ANOVA; ANOVA model: 1) Fixed effects: Sequence, Period, and Formulation; 2) Random effects: Volunteer (Sequence) and Residual; Ratio Geometric means T/R formulation = 90.03, 90% CI 2-sided [86.96 to 93.12], Standard Deviation 7.51 — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Time of Maximum Observed Concentration (Tmax)
Description: The time of maximum observed concentration (Tmax) is obtained directly from the plasma concentration curve of the drug by non-compartimental method. Tmax is of particular use in measuring bioavailability, by measuring the time at which the maximum concentration is achieved.
Time Frame: Collection points (hrs):0.00; 0.25; 0.50; 0.75; 1.00; 1.25; 1.50; 1.75; 2.00; 2.50; 3.00; 4.00; 5.00; 6.00; 8.00 evaluated in both periods: (Day 1 of Period 1 [Day 1 of study]; Day 1 of Period 2 [Day 15 of study])
Population: Entire Study Population
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 28 | 28
hr | 1.304 (0.468) | 1.482 (0.535)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.3390, Wilcoxon (Mann-Whitney); The non-parametric method included the following factors: Sequence, Formulation, Period, Formulation and Residual; Median Difference (Final Values) = 0.125, 90% CI 2-sided [-0.125 to 0.375]

5. Primary Outcome: Percentage of AUC0-inf That is Due to Extrapolation From the Time of the Last Measurable Concentration to Infinity (AUC%Extrapolation)
Description: The percentage of AUC0-inf that is due to extrapolation from Tlast to infinity (AUC%Extrapolation) is calculated by using the formula AUC_%extrapolation = 100*(AUC0-inf minus AUC0-t)/AUC0-inf. The function of this parameter is to provide information about what percentage of the theoretical curve (AUC0-inf) was possible to determine experimentally (AUC0-t) Therefore, on average, it is expected that the residual area (AUCextrapolation) is not greater than 20%.
Time Frame: as for outcome 4
Population: Entire Study Population
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 28 | 28
percentage | 1.303 (0.814) | 1.353 (0.743)

6. Primary Outcome: Terminal Half-life (T1/2_Kel)
Description: T1/2_Kel is calculated by using the formula T1/2_Kel = Ln(2)/Kel.T1/2 is of particular use in measuring bioavailability, by measuring the elimination of the product.
Time Frame: as for outcome 4
Population: Entire Study Population
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 28 | 28
hr | 1.085 (0.071) | 1.137 (0.155)

7. Primary Outcome: First-order Rate Constant Associated With the Terminal Portion of the Curve (Kel)
Description: This parameter is estimated via linear regression of time versus log concentration. It allows for the obtainment of estimates of T1/2 (T1/2=ln(2)/Kel) considering the schedule and the detection limits defined.
Time Frame: as for outcome 4
Population: Entire Study Population
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 28 | 28
1/hr | 0.641 (0.043) | 0.620 (0.079)

ADVERSE EVENTS:
Groups:
- Test Product in Period 1 and Reference Product in Period 2: Test product: Amoxicillin powder for oral suspension (Clamoxyl) 500 mg/5 mL in Period 1; followed by a 14-day washout period during which no medication was administered; followed by reference product; Amoxil 50 mg/5 mL in Period 2
- Reference Product in Period 1 and Test Product in Period 2: Reference product: Amoxil 500 mg/5 mL in Period 1; followed by a 14-day washout period during which no medication was administered; followed by test product: Clamoxyl 500 mg/5 mL in Period 2
Arm/Group | Test Product in Period 1 and Reference Product in Period 2 | Reference Product in Period 1 and Test Product in Period 2
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 10/14 | 4/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Product in Period 1 and Reference Product in Period 2 (N=14) | Reference Product in Period 1 and Test Product in Period 2 (N=14)
Headache (General disorders) | 3 | 0
Head throbbing (General disorders) | 0 | 1
Tension headache (General disorders) | 1 | 0
Urea increased (Renal and urinary disorders) | 0 | 1
Triglycerides increased (Blood and lymphatic system disorders) | 1 | 0
Glucose increased (Blood and lymphatic system disorders) | 1 | 0
Bilirubin total increased (Hepatobiliary disorders) | 0 | 1
Abnormal urine test results (Renal and urinary disorders) | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.